CLINICAL TRIAL: NCT01475162
Title: Phase I-II Study Using Tocilizumab for Treatment of Steroid Refractory Acute Graft-versus-Host Disease
Brief Title: Tocilizumab for Treatment of Steroid Refractory Acute Graft-versus-Host Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The DSMB felt the risks of the study now outweighed the potential benefits.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William R. Drobyski, MD, Professor of Medicine, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCW-PRO15904
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Acute Graft Versus Host Disease
Keywords: acute Graft versus Host Disease (aGVHD); steroid refractory acute Graft versus Host Disease (aGVHD); chronic Graft versus Host Disease (cGVHD); corticosteroids; allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tocilizumab (Experimental): Drug: Tocilizumab
  Other Names:
  Actemra
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks for three doses. After Day 56 doses may be decreased to 4mg/kg once every three weeks depending on GVHD response.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks for three doses. After Day 56 doses may be decreased to 4mg/kg once every three weeks depending on GVHD response.
  Other Names: Actemra

SUMMARY:
This trial designed to evaluate the toxicity and efficacy of tocilizumab in the treatment of steroid refractory acute graft versus host disease (GVHD).

DETAILED DESCRIPTION:
Patients who underwent an allogeneic hematopoietic stem cell transplantation, with biopsy proven GVHD, active acute GVHD requiring systemic immune suppressive therapy and that failed or did not respond to first line of therapy (corticosteroids ± other agent).

Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks. Patients with documented responses will continue to receive treatment at 8 mg/kg once every 3 weeks for at least two months (day 56). Patients that have some degree of response but without complete resolution of signs and symptoms of acute GVHD may continue to receive 8 mg/kg on a 3-week cycle until complete response is achieved or lack of further improvement. In patients who are beyond day 56 and whose GVHD has resolved, the dose of Tocilizumab will be reduced to 4 mg/kg every 3 weeks. Subsequent discontinuation of Tocilizumab will occur once patients are off other immune suppressive medications (including extracorporeal photopheresis, ECP) or are receiving sub therapeutic levels of immunosuppression (i.e., Tacrolimus (FK) levels <5 ng/mL) or prednisone dose <20 mg/day (or equivalent) and are free of acute GVHD signs or symptoms for at least one month.

Patients who fulfill criteria of progression of GVHD not in the setting of immunosuppressive taper, no response of GVHD or require initiation of other immune suppressive treatment for GVHD will have Tocilizumab discontinued.

Tocilizumab shall be discontinued and not re-instituted if any one of the following criteria is met. The patient will be taken off study drug therapy at that point, but still followed for primary and secondary study endpoints. A response assessment will be made at the time of therapy discontinuation and at subsequent defined study endpoints. The patient will not be replaced on study. Follow-up data will be required unless consent for data collection is withdrawn:

* Additional systemic GVHD therapy is added for disease progression or non-response
* Steroid dose is escalated to ≥ 2.5 mg/kg/day of prednisone (or methylprednisolone equivalent of 2 mg/kg/day) for GVHD progression or no response
* Development of toxicity that requires withholding of study medication for more then 14 days

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older who underwent an allogeneic hematopoietic stem cell transplantation.
* Patients are required to have biopsy proven GVHD.
* Patients must have active acute GVHD requiring systemic immune suppressive therapy and that failed or did not respond to first line of therapy.

  * First line therapy needs to be a minimum of corticosteroids, methylprednisolone of 1.6mg/kg/day or prednisone of 2mg/kg/day, alone or combined to other agent.
  * Failure of GVHD therapy is defined as flare of signs and symptoms of acute GVHD or progression of GVHD grade after at least 72 hours from starting therapy.
  * No response to GVHD treatment (corticosteroids ± other agent) after a minimum of 7 days of treatment.
* Patient must be able to give informed consent.

Exclusion Criteria:

* Intolerance or allergy to Tocilizumab
* Active uncontrolled infection requiring ongoing treatment with antifungals, antibiotics or anti-viral drugs.
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal.
* Liver enzymes: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3x upper limit of normal.
* Patients with severe sinusoidal obstruction syndrome who in the judgment of the treating physician are not expected to have normalized bilirubin by day 56 after enrollment.
* Serum bilirubin > 2x upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08-08 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2018-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William R Drobyski, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital/Medical College of Wisconsin-Clinical Cancer Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Drug: Tocilizumab Other Names: Actemra
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks for three doses. After Day 56 doses may be decreased to 4 mg/kg once every three weeks depending on graft versus host disease (GVHD) response.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 14
Completed | 0
Not Completed | 14
Not completed — Physician Decision | 1
Not completed — Death | 10
Not completed — Study closed for safety | 3

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab: Drug: Tocilizumab
  Other Names:
  Actemra
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks for three doses. After Day 56 doses may be decreased to 4mg/kg once every three weeks depending on GVHD response.
  Tocilizumab: Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks for three doses. After Day 56 doses may be decreased to 4mg/kg once every three weeks depending on GVHD response.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Complete or Partial Response at Day 56 After Administration of Tocilizumab
Description: Number of subjects achieving Center for International Blood and Marrow Transplant Research (CIBMTR) score of 0 (complete response); or achieving improvement in one or more organs involved in GVHD without progression in other organs (partial response). CIBMTR score of 0 means no evidence of rash or diarrhea and bilirubin less than 2.0 mg/dl. CIBMTR score of 4 means rash with bullae desquamation, lower gastrointestinal diarrhea more than 1,500 ml, and bilirubin greater than 15.1 mg/dl. Higher score means worse disease.
Time Frame: Day 56
Population: 6 of the thirteen subjects were not evaluable due to expiring prior to Day 56.
Measure: Count of Participants; unit: Participants
Groups:
- Tocilizumab: Drug: Tocilizumab Other Names: Actemra
  Tocilizumab will be administered intravenously at a dose of 8 mg/kg once every three weeks. Patients with documented responses will continue to receive treatment at 8 mg/kg once every 3 weeks for at least two months (day 56). Patients that have some degree of response but without complete resolution of signs and symptoms of acute GVHD may continue to receive 8 mg/kg on a 3-week cycle until complete response is achieved or lack of further improvement. In patients who are beyond day 56 and whose GVHD has resolved, the dose of Tocilizumab will be reduced to 4 mg/kg every 3 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Number of Patients With Partial, Mixed or no GVHD Responses
Description: Number of subjects achieving improvement in one or more organs involved in GVHD with or without deterioration in another organ (mixed or partial response, respectively); or having received additional immune suppressive therapy (no response).
Time Frame: Day 56
Population: Six subjects expired prior to day 56.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Participants | 2

3. Secondary Outcome: GVHD Flares
Description: Number of subjects exhibiting any progression requiring re-escalation of steroid dosing or initiation of additional topical or systemic therapy after achieving an initial complete or partial response prior to Day 90.
Time Frame: Day 90
Population: Six subjects expired prior to day 90.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Participants | 1

4. Secondary Outcome: Discontinuation of Immunosuppression
Description: Number of subjects for whom immunosuppressive therapy (corticosteroid, cyclosporine, tacrolimus, sirolimus, etc.) was discontinued. This will be evaluated at Day 56, Day 180 and Day 365.
Time Frame: Day 56, Day 180 and Day 365
Population: Six subjects expired prior to day 56.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Participants
  Day 56 | 0
  Day 180 | 0
  Day 365 | 1

5. Secondary Outcome: Overall Survival
Description: Number of subjects alive at one year.
Time Frame: 1 year
Population: For this analysis, all thirteen subjects meeting eligibility criteria were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 13
Participants | 3

6. Secondary Outcome: Number of Subjects Experiencing at Least One Serious Adverse Event or Grade 3 Non-serious Adverse Event
Description: Number of subjects experiencing at least one serious adverse event or adverse event of CTCAE grade 3, 4, or 5 at Day 56 following the initiation of tocilizumab therapy.
Time Frame: Day 56
Population: Six subjects expired prior to day 56.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
Participants | 7

7. Secondary Outcome: Disease-free Survival
Description: Number of subjects alive and not experiencing GVHD signs or symptoms at 6 and 12 months. At the six month time point, seven subjects had expired. At the 12 month time point, 10 subjects had expired.
Time Frame: 6 and 12 months
Population: For this analysis, all thirteen participants originally meeting eligibility criteria were included for evaluation of survival status. Living patients were evaluated for symptoms.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 13
Participants
  6 Month Timepoint: number analyzed (Participants) | 6
  6 Month Timepoint | 4
  12 Month Timepoint: number analyzed (Participants) | 3
  12 Month Timepoint | 3

8. Secondary Outcome: Non-relapse Mortality
Description: Number of subjects expiring from causes other than relapse of GVHD disease.
Time Frame: 6 months
Population: All thirteen subjects meeting the initial eligibility criteria were included for evaluation of survival status and cause of death.
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 13
Participants | 8

ADVERSE EVENTS:
Time Frame: An average of one year.
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 10/13
Serious Adverse Events (participants affected / at risk) | 13/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=13)
Elevated alanine aminotransferase Grade 3 (Investigations) | 1 (1)
Adult respiratory distress syndrome Grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea Grade 3 (Gastrointestinal disorders) | 1 (1)
Diarrhea Grade 4 (Gastrointestinal disorders) | 1 (1)
Sepsis Grade 5 (Infections and infestations) | 3 (3)
Sepsis Grade 4 (Infections and infestations) | 3 (3)
Presyncope Grade 1 (Nervous system disorders) | 1 (1)
Bronchial infection Grade 3 (Infections and infestations) | 1 (1)
Enterocolitis Grade 3 (Gastrointestinal disorders) | 1 (1)
Pneumothorax Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multi-organ failure Grade 5 (General disorders) | 1 (1)
Blood and lymphatic system disorders - Other Grade 5 (Blood and lymphatic system disorders) | 1 (1)
Adult respiratory distress syndrome Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-02-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT01475162/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT01475162/Prot_SAP_001.pdf